CLINICAL TRIAL: NCT03828006
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Clinical Trial to Demonstrate the Efficacy of a Dietary Supplement in Decreasing Cardiovascular Risk
Brief Title: Clinical Trial to Demonstrate the Efficacy of a Dietary Supplement in Decreasing Cardiovascular Risk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bioksan (Industry)
Collaborators: Analysis and Research Network, S.L (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BIO-LIP-01-18
Record Dates: First submitted 2019-01-10; First posted 2019-02-04 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-07

CONDITIONS: Low-Moderate Hypercholesterolemia
MeSH Terms: interventions — red yeast rice

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): One tablet per day through oral administration of a dietary supplement containing red rice yeast as the main active ingredient
  Interventions: Dietary Supplement: Red Rice Yeast
- Placebo Group (Placebo Comparator): One tablet per day of placebo.
  Interventions: Other: Placebo Group

INTERVENTIONS:
Dietary Supplement: Red Rice Yeast — Participants will take one tablet per day of a dietary supplement based on red rice yeas for a period of six months
  Arms: Active Group
Other: Placebo Group — Participants of this group will take one tablet of placebo per day for a period of six months
  Arms: Placebo Group

SUMMARY:
This clinical trial seeks to verify the efficacy of a red rice yeast dietary supplement in the decrease of cardiovascular risk, by assessing variables related with cardiovascular risk as levels of cholesterol, triglycerides and transaminases among other, in two groups of participants that will be taking either the dietary supplement or a placebo during a six months period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old or older
* Body Mass Index (BMI) between 18.5 y 29.9.
* LDL-c levels between 100mg/dL and 160mg/dL
* 10 year estimated cardiovascular risk assessed by the ASCVD less than 20%
* Accepts to participate and sings Informed Consent.

Exclusion Criteria:

* Patients with history of cardiovascular diseases.
* Patients with secondary hyperlipidemia caused by diabetes mellitus, or kidney, liver or thyroid diseases.
* Patients with muscle diseases
* Patients undergoing pharmacological treatment with any of the following: lipid lowering agents, antifungal, macrolides, or hormone replacement therapy in progress or during the last 2 months.
* Patients with proven intolerance with the components present in the dietary supplement.
* Patients with any other concomitant disease that to the researcher's criteria are not susceptible to participate in the study.
* Woman that are pregnant, in breastfeeding period or with a possibility of starting a pregnancy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Systematic Coronary Risk Evaluation (SCORE) | Changes in the score from the baseline, at 3 and 6 months.
  This scale estimates the 10 year risk of fatal CVD.
  The risk is estimated with a High & Low cardiovascular Risk Charts based on gender, age, total cholesterol, systolic blood pressure and smoking status, with relative risk chart, qualifiers and instructions. High risk or low risk table depends on whether the person lives in a high or low risk country.
  There possible scores goes from 0 to 47 in the high risk table, and 0 to 26 in the low risk table. Where lower values represent lower risk and higher values higher risk.
Arteriosclerotic Cardiovascular Disease Algorithm (ASCVD) | Changes in the score from the baseline, at 3 and 6 months.
  Calculates 10-year risk of heart disease or stroke using the ASCVD algorithm published in 2013 American College of Cardiology/American Heart Association (ACC/AHA) Guidelines on de Assessment of Cardiovascular Risk.
Registre Gironi del Cor (REGICOR) | Changes in the score from the baseline, at 3 and 6 months.
  The scale measures the probability of having cardiovascular disease in 10 years.
  The probability is estimated with age, sex, smoking status, diabetic or not, total Cholesterol (mg/dl), HDL cholesterol (mg/dl), systolic blood pressure (mmHg) and diastolic blood pressure (mmHg).
  Possible risk values are divided in 5 categories: low <5%, moderate 6-9%, medium 10-19%, high 20-38%, very high >39%

SECONDARY OUTCOMES:
Changes in LDL cholesterol levels in blood | Changes in the cholesterol levels from the baseline, at 3 and 6 months.
  LDL in blood measured in mg/dL Measurements will be taken at basal visit, at 3 months and at 6 months after the start of the dietary supplement/placebo intake.
Changes in HDL cholesterol levels in blood | Changes in the cholesterol levels from the baseline, at 3 and 6 months.
  HDL cholesterol will be measured in mg/dl Measurements will be taken at basal visit, at 3 months and at 6 months after the start of the dietary supplement/placebo intake.
Changes in triglycerides levels in blood | Changes in the triglyceride levels from the baseline, at 3 and 6 months.
  Triglycerides will be measured in mg/dl Measurements will be taken at basal visit, at 3 months and at 6 months after the start of the dietary supplement/placebo intake.
Changes in lipoprotein levels in blood | Changes in the lipoprotein levels from the baseline, at 3 and 6 months.
  Lipoproteins will be measured in mg/dl Measurements will be taken at basal visit, at 3 months and at 6 months after the start of the dietary supplement/placebo intake.
Levels of glycosylated hemoglobin in blood | Changes in the lipoprotein levels from the baseline, at 3 and 6 months.
  Glycosylated Hemoglobin (HbA1c) will be measured as % in blood Measurements will be taken at basal visit, at 3 months and at 6 months after the start of the dietary supplement/placebo intake.
Alanine Transaminase (ALT) levels | Changes in the lipoprotein levels from the baseline, at 3 and 6 months.
  Levels of ALT Transaminase measured in IU/L. Measurements will be taken at basal visit, at 3 months and at 6 months after the start of the dietary supplement/placebo intake.
Adverse Events | Through study completion, an average of 9 months
  Number of adverse events.
Therapeutic adherence | At the 6 month visit
  Data will be collected by the investigator at participant visits with a unique question about percentage of intake. It will be considered a good compliance if the 80% of the medication has been taken.
Morisky-Green scale | At the 6 month visit
  The Morisky-Green scale measures treatment adherence with four yes or no questions.
  In which yes punctuates 0 and no punctuates 1.
  Possible result values goes from 0 to 4, being 0 less adherence and 4 more adherence.
Recount of returned product | At the 6 month visit
  The number of returned product will be counted

CONTACTS AND LOCATIONS:
Locations (3):
- Spain (3):
  - Hospitales San Roque, Las Palmas de Gran Canaria, Canary Islands
  - Hospital Universitari de Bellvitge, Barcelona, Catalonia
  - Hospital General Universitari de València, Valencia